CLINICAL TRIAL: NCT01653964
Title: Evaluation of Half-Dose Molecular Breast Imaging With Wide Beam Reconstruction Processing
Acronym: Split-Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Friends for an Earlier Breast Cancer Test (Unknown)
Responsible Party: Principal Investigator, Carrie Hruska, Prinicipal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-004437
Record Dates: First submitted 2012-07-24; First posted 2012-07-31 (Estimated); Results first posted 2017-09-18 (Actual); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: suspicious; lesion; breast; cancer; screening; mammogram; negative
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Molecular breast imaging (Experimental): Molecular Breast Imaging at 4 mCi dose and at 8 mCi dose, consecutively.
  Interventions: Diagnostic Test: Molecular breast imaging

INTERVENTIONS:
Diagnostic Test: Molecular breast imaging — Molecular breast imaging performed with injection of Tc-99m sestamibi and a dedicated gamma camera (Luma Gem, Gamma Medica)

SUMMARY:
The primary objective of this work is to determine if half-dose Molecular Breast Imaging (MBI) performed with 4 mCi Tc-99m sestamibi with or without Wide Beam Reconstruction applied can achieve image quality and diagnostic accuracy non-inferior to that of standard MBI performed with 8 millicurie (mCi) Tc-99m sestamibi.

DETAILED DESCRIPTION:
Recent implementation of dose reduction strategies for Molecular Breast Imaging now allow performance of MBI at an administered dose of 8 mCi Tc-99m sestamibi, which is reduced from the previously used doses of 20-30 mCi. In order to safely introduce MBI as a screening modality, we aim to perform MBI using 4 mCi Tc-99m sestamibi. An image processing algorithm called Wide Beam Reconstruction (WBR) has been tailored for MBI technology with the goal of allowing either the current administered dose or current acquisition time to be reduced by half.

ELIGIBILITY:
Inclusion Criteria:

Subgroup 1, Patients with breast lesions:

-At least one breast lesion detected by mammogram, ultrasound or breast MRI that measures < 20 mm in greatest dimension, presents as a mass, is considered suspicious or highly suggestive of malignancy according to the Breast Imaging Reporting and Data System Atlas criteria (BIRADS 4 or 5), and is scheduled for core-needle biopsy or surgical biopsy.

OR

-At least one breast lesion that measures between > 10 mm but < 20 mm in greatest dimension, presents as a mass, is biopsy-proven as malignant, and is scheduled for surgical resection.

AND

* Age > 40 years
* Negative pregnancy test, postmenopausal, or surgically sterilized

Subgroup 2, Patients without known breast lesions:

* Negative screening mammogram performed at Mayo Clinic Rochester within 15 months prior to performance of study MBI
* No signs or symptoms of breast disease
* Age > 40 years
* Negative pregnancy test, postmenopausal, or surgically sterilized

Exclusion Criteria:

* Vacuum-assisted or excisional biopsy has been performed prior to the study MBI. Reason: these types of biopsies are more likely to remove all of the tumor
* MBI is performed after biopsy and neo-adjuvant chemotherapy is planned prior to surgery. Reason: true tumor size will not be able to be ascertained from the final pathology findings
* Breast implants. Reason: cases with breast implants will be easily identifiable on blinded interpretation to take place at the study end
* Suspected that breasts will not fit in the MBI field of view. Reason: cases that require tiled views or additional views will be easily identifiable on blinded interpretation to take place at the study end
* Only one breast remaining. Reason: unilateral cases will be easily identifiable on blinded interpretation to take place at the study end; injection timing is designed for bilateral views
* Pregnancy test (if necessary) is not negative, or the patient is unable to complete the pregnancy test
* Physically unable to sit upright and still remain still during two consecutive MBI studies over the course of a 2-hour period.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carrie B Hruska, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic News — http://newsblog.mayoclinic.org/2008/09/03/breast-cancer-molecular-breast-imaging-mammography/
- See also: Mayo Clinic You Tube Channel — http://www.youtube.com/watch?v=DOQBLe8MdH0

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 83 subjects were enrolled (consented) but 1 subject was found not to meet eligibility criteria, so did not participate in the study.
Groups:
- Molecular Breast Imaging: Molecular breast imaging performed after injection of 4 mCi Tc-99m sestamibi and again after 8 millicurie (mCi) Tc-99m sestamibi.
Period: Overall Study
Arm/Group | Molecular Breast Imaging
Started | 82
Completed | 82
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Molecular Breast Imaging
Number analyzed (Participants) | 82
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 82
  More than one race | 0
  Unknown or Not Reported | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 82

OUTCOME MEASURES:

1. Primary Outcome: Compare the Diagnostic Accuracy of 8 mCi Molecular Breast Imaging (MBI) With 4 mCi MBI.
Time Frame: At time of study (within 2 days after exam) and when enrollment has been reached (approximately 24 months)
Population: Of 82 patients recruited to the study (prior to breast biopsy), 34 had a histologically-proven diagnosis of breast cancer.
Measure: Number; unit: cancers detected
Groups:
- Molecular Breast Imaging: Molecular breast imaging performed after injection of 4 mCi Tc-99m sestamibi and again after 8 mCi Tc-99m sestamibi.
Arm/Group | Molecular Breast Imaging
Number analyzed (Participants) | 34
cancers detected
  8 mCi | 30
  4 mCi | 29

ADVERSE EVENTS:
Time Frame: Day of study participation
Arm/Group | Molecular Breast Imaging
All-Cause Mortality (participants affected / at risk) | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82
Other Adverse Events (participants affected / at risk) | 0/82

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No